CLINICAL TRIAL: NCT00005684
Title: Oral Anticoagulant Therapy for Venous Thrombosis - SCOR in Thrombosis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4108; P50HL054502 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-02

CONDITIONS: Venous Thrombosis; Cardiovascular Diseases; Venous Thromboembolism
MeSH Terms: conditions — Venous Thrombosis; Cardiovascular Diseases; Venous Thromboembolism | interventions — Warfarin; Heparin

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Drug: warfarin
Drug: heparin

SUMMARY:
To perform a randomized clinical trial comparing continuing one month of treatment with heparin in patients with deep venous thrombosis to standard care using heparin for five days and oral warfarin for three months.

DETAILED DESCRIPTION:
BACKGROUND:

The study, a subproject within a SCOR in Thrombosis, should help to improve the long-term clinical outcome of patients with proximal deep-vein thrombosis (popliteal, femoral or iliac vein thrombosis) by improving their survival and reducing morbidity from recurrent thromboembolic events, and should help to determine if one or more specific biochemical measures, including antiphospholipid antibodies and activated factor VII, will define a subset of patients at increased risk of recurrent venous thromboembolism.

The study is part of a SCOR in Hemostatic and Thrombotic Diseases, the RFA for which was released by the NHLBI in April 1994.

DESIGN NARRATIVE:

Warfarin Trial

A multicenter, randomized clinical trial was conducted from March 1996 through January 2001 comparing warfarin therapy for three years to warfarin therapy for three months. The study was performed at thirteen participating hospitals in Oklahoma. The 600 hundred patients were recruited, randomized to either warfarin therapy for three years or warfarin therapy for three months and followed for at least three years. The primary outcome measure was total mortality. Secondary outcome measures included vascular death, objectively documented recurrent venous thromboembolism, and bleeding complications (major and minor). Additional specific aims included: determining the prevalence of antiphospholipid antibodies, antithrombomodulin antibodies, and activated protein C resistance in consecutive patients with proximal-vein thrombosis; determining if these measures, and/or the level of activated factor VII were associated with an increased risk of recurrent venous thromboembolic events, and if so, whether these events were reduced by continuing long term warfarin treatment. These latter specific aims were achieved by performing the laboratory parameters concurrently in patients entered into the clinical trial, and relating these measures to the clinical outcomes on long-term follow-up.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-03; Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Raskob — Oklahoma Medical Research Foundation